CLINICAL TRIAL: NCT04046159
Title: Radiotherapy Versus Low-Dose Tamoxifen Following Breast Conserving Surgery for Low-Risk and Estrogen Receptor-Positive Ductal Carcinoma in Situ of Breast: an International Open-label Randomized Non-inferiority Trial
Brief Title: Radiotherapy Versus Low-Dose Tamoxifen Following Breast Conserving Surgery for Low-Risk Breast Ductal Carcinoma in Situ
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Tri-Service General Hospital (Other); Koo Foundation Sun Yat-Sen Cancer Center (Other); Kaohsiung Medical University (Other); Kyoto University (Other); Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201902048MINC
Record Dates: First submitted 2019-07-07; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-04

CONDITIONS: Breast Ductal Carcinoma in Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: Non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy arm (Active Comparator): Radiotherapy for ipsilateral whole breast with 50 Gy/25 fractions or 40.05 Gy/15 fractions
  Interventions: Radiation: Whole breast radiotherapy
- Tamoxifen arm (Experimental): Tamoxifen 5 mg QD for 10 years
  Interventions: Drug: Low-dose tamoxifen

INTERVENTIONS:
Drug: Low-dose tamoxifen — Low-dose tamoxifen is not inferior than radiotherapy in decreasing ipsilateral breast tumor recurrence and side effect
  Other Names: LDT
  Arms: Tamoxifen arm
Radiation: Whole breast radiotherapy — Ipsilateral breast tumor recurrence and side effect
  Other Names: WBRT
  Arms: Radiotherapy arm

SUMMARY:
Although the results obtained from ECOG E5194 cohort 1 (criteria: mammographically detected low- or intermediate-grade DCIS, measuring less than 2.5 cm with margins ≥ 3 mm) and RTOG 9804 trial (the same enrolled clinicopathological features to cohort 1 of ECOG E5194 trial) demonstrated that the 7-year ipsilateral breast tumor recurrence (IBTR) ranged from 5.6% to 10.5% for low-risk ductal carcinoma in situ (DCIS) patients, the aforementioned two studies included a proportional patients who had young age and negative estrogen receptor (ER) status tumor. Previous studies and our studies revealed that age < 40 years and ER-negative status in tumor were independent prognostic factor for recurrence of breast DCIS irrespective of tumor characteristics. The UK/ANZ randomized trial, enrolling high-risk and low-risk clinicopathologic features of DCIS, demonstrated that a benefit of tamoxifen in terms of reducing the IBTR is observed in the BCS alone group but not found in the BCS plus RT group. A recent published randomized trial showed that tamoxifen at the dose of 5 mg/day for 3 years.

Based on the aforementioned results, we hypothesized that the administration of tamoxifen is not inferior than the prescription of RT in terms of reducing the IBTR for DCIS patients who had age more than 40 years, the pathological features meeting the ECOG E5194 cohort 1 criteria, and positive ER status in tumors. To approve the hypothesis, we will design a randomized non-inferiority trial to assess whether the effect of administration of tamoxfien (5 mg per day) for 10 years following BCS is not inferior in terms of reducing IBTR when comparing RT following BCS for patients who had low-risk clinicopathologic features (age more than 40 years and ECOG E5194 cohort 1 criteria) and positive-ER status of breast DCIS.

DETAILED DESCRIPTION:
[Background] Radiotherapy (RT) following breast conserving surgery (BCS) is commonly used in ductal carcinoma in situ (DCIS) of breast to decrease local recurrence. Previous retrospective studies suggested that a substantial proportional of low-risk DCIS patients who underwent BCS alone will not develop a subsequent invasive breast cancer over time.

To further identify a population of patients with low-risk DCIS in whom adjuvant RT could be safely omitted, two prospective trials and one randomized trial have been published the ipsilateral breast tumor recurrence (IBTR) rate in patients with low-risk breast DCIS, including smaller size, larger margin width, and lower grade. The 5-year IBTR rate in Dana Farber/Harvard Cancer Institute (low to intermediate grade disease and a margin width of 10 mm) was 12% for breast DCIS patients who underwent BCS alone. The Eastern Cooperative Oncology Group (ECOG) E5194 reported a 12-year IBTR rate of 14.4% (7-year IBTR rate, 10.5%) for patients with low-risk DCIS (cohort 1 criteria: mammographically detected low- or intermediate-grade DCIS, measuring less than 2.5 cm with margins ≥ 3 mm) who underwent BCS alone. The risk for DCIS and invasive cancer increased steadily over time, without any plateau.

Another randomized trial, Radiation Therapy Oncology Group (RTOG) 9804, showed the IBTR rates from that at 5 years (3.5%) to that at 7 years (6.7%) in post-BCS patients with low-risk breast DCIS (similar criteria of ECOG E5194 trial, cohort 1) who did not receive RT. In contrast, the 7-year IBTR rate was low (0.9%) for patients who underwent BCS and received RT in RTOG 9804 trial. Our retrospective study showed that the 7-year IBTR rate was 5.6% in breast DCIS patients who had criteria of cohort 1 of ECOG E5194 trial and underwent BCS alone. Taken together, two prospective clinical trials and our retrospective study disclosed that the 7-year IBTR for BCS alone group (no RT) ranged from 5.6% to 10.5%, even if patients whose clinicopathologic features met the criteria of ECOG E5194 cohort 1. These results suggest that RT following BCS is indicated for these patients who have low-risk breast DCIS.

Another randomized trial, UK/ANZ [UK, Australia, and New Zealand] DCIS trial], including high-risk and low-risk breast DCIS patients, demonstrated a significant benefit of tamoxifen (20 mg every day for 5 years) in terms of reducing the ipsilateral (Hazard ratio [HR], 0·77; 95% confidence interval [CI], 0·59-0·98; P = 0·04) and contralateral breast events (HR, 0·27; 95% CI, 0·12-0·59; P = 0·001) in the BCS alone group, and this benefit of tamoxifen was not observed in the BCS plus RT group for ipsilateral events (HR, 0·93; 95%, 0·50-1·75; P = 0·8). These findings suggest that even if patients with low-risk clinicopatholgical features of DCIS (relatively low-risk of IBTR), the addition of tamoxifen in patients who had received RT may not reduce IBTR than those receiving RT alone. However, the estrogen receptor (ER) status among the patients with DCIS enrolled in the aforementioned three prospective randomized trials (ECOG E5194 trial, RT9804 trial, and UK/ANZ trial) was initially unknown.

In a retrospective analysis of the relationship between ER status and response to tamoxifen in 732 patients (41%) who comprised the original NSABP B-24 population (76% positive for ER), the significant effect of tamoxifen in reducing ipsilateral and contralateral breast events was demonstrated in ER-positive DCIS but not in ER-negative tumors. Our retrospective study also showed that age < 40 years and negative ER status in tumors were closely associated with the higher IBTR rate. Among our patients with cohort 1 criteria of ECOG E519 study, the 7-year IBTR rate for ER-positive group and ER-negative group was 5.0% and 8.0%, respectively.

[Rationale] Although the results obtained from ECOG E5194 (cohort 1) and RTOG 9804 trial (the same enrolled clinicopathological features to cohort 1 of ECOG E5194 trial) demonstrated that the 7-year IBTR ranged from 5.6% to 10.5% for low-risk DCIS patients, the aforementioned two studies included a proportional patients who had young age and negative ER status tumor. Previous studies and our studies revealed that age < 40 years and ER-negative status in tumor were independent prognostic factor for recurrence of breast DCIS irrespective of tumor characteristics.

The UK/ANZ randomized trial, enrolling high-risk and low-risk clinicopathologic features of DCIS, demonstrated that a benefit of tamoxifen in terms of reducing the IBTR is observed in the BCS alone group but not found in the BCS plus RT group. In a recent published data of a randomized trial of comparing low-dose tamoxifen (5 mg QD) for 3 years with placebo in prevention of recurrence of women with hormone-positive DCIS or lobular carcinoma in situ, low-dose tamoxifen was demonstrated to significantly decrease local recurrence when compared with placebo arm. These findings indicate that tamoxifen at the dose of 5 mg/day can decrease the incidence of recurrence in women with operated hormone sensitive DCIS with a limited toxicity. However, the effect of the administration of low-dose tamoxifen is similar to the RT effect in terms of reducing IBTR for patients who had the criteria of ECOG E5194 cohort 1 and positive ER status remains unclear.

[Hypotheses] Based on the aforementioned results, we hypothesized that the administration of tamoxifen is not inferior than the prescription of RT in terms of reducing the IBTR for DCIS patients who had age more than 40 years, the pathological features meeting the ECOG E5194 cohort 1 criteria, and positive ER status in tumors.

To approve the hypothesis, we will design a randomized non-inferiority trial to assess whether the effect of administration of tamoxfien (5 mg per day) for 10 years following BCS is not inferior in terms of reducing IBTR when comparing RT following BCS for patients who had low-risk clinicopathologic features and positive-ER status of breast DCIS.

[Study Design] We will design a randomized non-inferiority trial to assess whether the effect of administration of tamoxfien (5 mg) for 10 years following BCS is not inferior in terms of reducing IBTR when comparing RT (in terms of 50 Gy in 25 fractions or 40.05 Gy in 15 fractions) following BCS for patients who had age more than and equal 40 years, low-risk clinicopathological features (ECOG E5194 cohort 1 criteria), and positive-ER status of breast DCIS.

ELIGIBILITY:
Inclusion Criteria:

1. Women
2. New histologically diagnosed breast ductal carcinoma in situ (DCIS).
3. Age ≥ 40 years
4. Low risks of BRCA (breast cancer)1 and BRCA2: Manchester Score < 10
5. The DCIS must be detected by mammogram and must be unicentric, and no-mass lesion.
6. Status post breast conserving surgery
7. Pathological characteristics (all characteristics) 7.1 Lesions ≤ 2.5 cm in greatest dimension on pathologic specimen (use the largest measured size from the pathology report to obtain the required measurement of ≤ 2.5 cm).

   7.2 Must be classified as low or intermediate nuclear grade DCIS but without comedo necrosis according to Pathologic Guidelines (section 9.2.2) 7.3 Margins as assessed by the ink method will be 3 mm or greater. 7.4 Must be estrogen receptor (ER)-positive DCIS, ER percentage must be ≥10%
8. Clinically node negative.

Exclusion Criteria:

1. Known BRCA1 or BRCA2 mutation
2. Age < 40 years
3. Women whose DCIS is palpable at the time of diagnosis, or multi-centric (mammography), or mass (mammography), or who have bloody nipple discharge.
4. Pathological characteristics 4.1 Lesions measuring greater than 2.5 cm in greatest dimension on pathologic specimen.

   4.2.High-grade lesions or low to intermediate grade with comedo necrosis as classified by the Guidelines.

   4.3. Margins as assessed by the ink method will be less than 3 mm. 4.4. ER-negative DCIS or ER-positive percentage < 10% in tumor cells
5. Post-mastectomy patients
6. Prior diagnosis of neoplasm within 5 years, except cervical intraepithelial neoplasia type 1 (CIN1) or localized non-melanomatous skin cancer.
7. Evidence of clinically significant cardiac disease, as defined by cardiac disease (New York Cardiac disease grade II), history of myocardial infarction, cerebral stroke, unstable arrhythmia, and unstable angina pectoris within 12 months before study entry.
8. Pregnant or lactating status.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 810 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Breast tumor recurrence | through study completion, an average of 1 year
  Ispilateral, regional recurrence, contralateral recurrence, and distant recurrence [DCIS or invasive cancer event]

SECONDARY OUTCOMES:
The overall survival | through study completion, an average of 1 year
  Overall survival
Adverse effects | through study completion, an average of 1 year
  Adverse effects of radiotherapy and tamoxifen

CONTACTS AND LOCATIONS:
Overall Officials: Chiun-Sheng Huang, MD, PhD, MPH, Principal Investigator — Department of Surgery, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Share participant data
Supporting Information: Study Protocol, CSR
Time Frame: 5 years after completion of study
Access Criteria: Will be available after contacting with Principle investigators

REFERENCES:
- [Derived] Kuo SH, Tseng LM, Chen ST, Sagara Y, Chang YC, Yeh HT, Kuo YL, Hung CC, Lu TP, Lee YH, Toi M, Huang CS. Radiotherapy versus low-dose tamoxifen following breast-conserving surgery for low-risk and estrogen receptor-positive breast ductal carcinoma in situ: an international open-label randomized non-inferiority trial (TBCC-ARO DCIS Trial). BMC Cancer. 2023 Sep 14;23(1):865. doi: 10.1186/s12885-023-11291-6. PMID 37710198